CLINICAL TRIAL: NCT07177638
Title: A Community-based Educational Initiative to Raise Awareness of Melanoma and Other Skin Cancers: Pilot Proof of Concept Study
Brief Title: A Community-based Educational Initiative to Raise Awareness of Melanoma and Other Skin Cancers.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-00625
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Skin Cancer
Keywords: Melanoma; Basal Cell Carcinoma; Squamous Cell Carcinoma; Education; South Brooklyn
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults from Bensonhurst County in Brooklyn, New York (Experimental): Participants will complete a pre-study survey and then take part in the educational session; follow-up visits to assess the impact of the intervention on participant knowledge and skin self-examination behaviors at will be held at 3 weeks, 3 months, 6 months, and 12 months. Participants will also complete a post-study survey at Month 12.
  Interventions: Behavioral: Education Sessions to Improve Melanoma Knowledge and Awareness

INTERVENTIONS:
Behavioral: Education Sessions to Improve Melanoma Knowledge and Awareness — Community based educational seminar led by a community health worker with follow-up questionnaires to assess knowledge retention and behavioral change.

SUMMARY:
This is a pilot study of a community- based melanoma educational intervention in Bensonhurst, Brooklyn conducted in-person by a community-health worker employed by the Perlmutter Cancer Center. Sample size will be around 35 participants. The participants will complete a pre-study survey and then take part in the educational session. There will be follow up study visits to assess the impact of the intervention on participant knowledge and skin self-examination behaviors at 3 weeks, 3 months, 6 months, and 12 months. At the 12-month mark, the participants will also complete a post-study survey.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Individuals who understand and speak either English or Russian
* Willingness and ability to consent and participate in the study

Exclusion Criteria:

* Under 18 years of age
* Individuals who do not understand and speak either English or Russian
* Individuals who participated in the focus group portion of a related study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Change in Melanoma Knowledge as Assessed by Questionnaire | Baseline, Immediately Post-Educational Session (Day 1)
  Melanoma knowledge/awareness will be assessed using a study questionnaire. Each item is multiple choice with 1 correct answer: the total score is the percentage of correct responses and ranges from 0-100%.
Change in Melanoma Knowledge as Assessed by Questionnaire | Baseline, Week 3 Post-Intervention
  Melanoma knowledge/awareness will be assessed using a study questionnaire. Each item is multiple choice with 1 correct answer: the total score is the percentage of correct responses and ranges from 0-100%.

SECONDARY OUTCOMES:
Change in Melanoma Knowledge as Assessed by Questionnaire | Month 3 Post-Intervention, Month 6 Post-Intervention
  Melanoma knowledge/awareness will be assessed using a study questionnaire. Each item is multiple choice with 1 correct answer: the total score is the percentage of correct responses and ranges from 0-100%.
Change in Melanoma Knowledge as Assessed by Questionnaire | Month 3 Post-Intervention, Month 12 Post-Intervention
  Melanoma knowledge/awareness will be assessed using a study questionnaire. Each item is multiple choice with 1 correct answer: the total score is the percentage of correct responses and ranges from 0-100%.
Change in Number of Self-Skin Examinations | Month 3 Post-Intervention, Month 6 Post-Intervention
  Assessed via survey.
Change in Number of Self-Skin Examinations | Month 3 Post-Intervention, Month 12 Post-Intervention
  Assessed via survey.

CONTACTS AND LOCATIONS:
Overall Officials: David Polsky, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- Jewish Community House of Bensonhurst, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: david.polsky@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to david.polsky@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.